CLINICAL TRIAL: NCT03569514
Title: An Observational Clinical Study of AIGIV Use in Sporadic Cases of Systemic Anthrax
Brief Title: Observational Study Evaluating Clinical Benefit and Safety of AIGIV (ANTHRASIL®) in Patients With Systemic Anthrax
Status: Not yet recruiting | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AX-003B
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anthrax
Keywords: Anthrax; Bacillus anthracis; Bacterial infection; AIGIV; Anthrax immune globulin; Anti toxin; Polyclonal antibodies
MeSH Terms: conditions — Anthrax; Bacterial Infections | interventions — Anthrax Immune Globulin Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AIGIV: Anthrax patients who have been administered AIGIV (ANTHRASIL®) as per licensed US prescribing information.
  Interventions: Drug: AIGIV

INTERVENTIONS:
Drug: AIGIV — Anthrax Immune Globulin Intravenous (Human)
  Other Names: ANTHRASIL®

SUMMARY:
This study will evaluate safety and clinical benefit of AIGIV used for treatment of patients with systemic anthrax. The study is designed to collect information on safety, clinical benefit (such as extent of anthrax illness and survival) and serum concentrations of AIGIV (for AIGIV pharmacokinetics) and anthrax toxins from sporadic cases of systemic anthrax patients treated with AIGIV.

DETAILED DESCRIPTION:
This study is a post-marketing requirement from the FDA to evaluate safety and clinical benefit of AIGIV administered to systemic anthrax patients as part of their medical care after exposure to Bacillus anthracis (anthrax exposure can be via inhalation, ingestion, injection). Study information (i.e. data on safety and clinical benefit evaluation of AIGIV up to Day 30 following administration) and patient samples (for assessment of AIGIV pharmacokinetics and anthrax toxin levels) will be collected (up to Day 7 following AIGIV administration) prospectively to the extent possible; however, in some cases data may be collected retrospectively (including scavenged patient samples for assessment of serum AIGIV concentration and anthrax toxin levels). Therefore, both prospective and retrospective data collection are allowed in this study to maximize the amount of information obtained from systemic anthrax patients who have been treated with AIGIV.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected systemic anthrax patients in the USA or other jurisdictions (if feasible) treated with AIGIV provided by the Centers for Disease Control and Prevention (CDC).
* Systemic anthrax defined as a clinically compatible case of gastrointestinal, injectional, or inhalational anthrax; anthrax meningitis or bacteremia; or cutaneous anthrax with systemic effects (i.e. tachycardia, tachypnea, hypotension, hyperthermia, hypothermia, leukocytosis) or with lesions that involve the head, neck or upper torso, or are large, bullous, multiple, or surrounded by significant edema PLUS confirmation by one of the following:

Epidemiologically linked to a documented anthrax environmental exposure. Laboratory confirmation by isolation of B. anthracis from an affected tissue or site.

Demonstration of B. anthracis antigens in tissues by immunohistochemical staining using both B. anthracis cell wall and capsule monoclonal antibodies.

Evidence of B. anthracis DNA; for example, by polymerase chain reaction (PCR) in specimens collected from a normally sterile site (such as blood or cerebrospinal fluid (CSF)) or lesion of other affected tissue(s) (skin, pulmonary, reticuloendothelial, or gastrointestinal).

QuickELISA™ Anthrax-PA kit manufactured by Immunetics, Inc. for detection of anti-PA antibodies in serum, plasma, and pleural/ascitic fluid.

RedLine Alert™ test manufactured by Tetracore, Inc., for identification of B. anthracis colonies.

* Informed consent/assent (as applicable).

Exclusion Criteria:

* There are no exclusion criteria for subjects enrolling in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anthrax patients who have received AIGIV.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-11-30 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of AIGIV clinical benefit by overall mortality rate | Up to Day 30
  Mortality rate (incidence of death) in patients with confirmed diagnosis of systemic anthrax treated with AIGIV

SECONDARY OUTCOMES:
Assessment of AIGIV safety by incidence of serious adverse drug reactions and serious suspected adverse drug reactions | Up to Day 30
  Combined incidence of serious adverse drug reactions (i.e. serious adverse events related to AIGIV administration) and serious suspected adverse drug reactions (i.e. serious adverse events that occur during or within 24 hours following AIGIV administration) in individuals treated with AIGIV

OTHER OUTCOMES:
Cause-specific mortality rate | Up to Day 30
  Number of deaths assigned to a specific cause in patients with confirmed diagnosis of systemic anthrax treated with AIGIV
Mortality rate stratified by number of AIGIV doses administered | Up to Day 30
  Number of deaths stratified by number of AIGIV doses (single versus multiple doses) in patients with confirmed diagnosis of systemic anthrax treated with AIGIV
Mortality rate stratified by AIGIV treatment time from symptom onset | Up to Day 30
  Number of deaths stratified by AIGIV treatment time from symptom onset (early versus late onset of symptoms) in patients with confirmed diagnosis of systemic anthrax
Mortality rate stratified by acute physiologic assessment and chronic health evaluation (APACHE) II score at baseline | Up to Day 30
  Number of deaths stratified by APACHE II score at baseline in patients with confirmed diagnosis of systemic anthrax treated with AIGIV
Duration of hospitalization | Up to Day 30
  Length of hospitalization in patients with confirmed diagnosis of systemic anthrax treated with AIGIV
Duration of intensive care unit (ICU) hospitalization | Up to Day 30
  Length of ICU stay in patients with confirmed diagnosis of systemic anthrax treated with AIGIV
Incidence of ICU hospitalization | Up to Day 30
  Number of patients with confirmed diagnosis of systemic anthrax treated with AIGIV admitted to ICU
Duration of mechanical ventilation | Up to Day 30
  Length of mechanical ventilation in patients with confirmed diagnosis of systemic anthrax treated with AIGIV
Evaluation of sequential organ failure assessment (SOFA) score | Up to Day 14
  Increase in sequential organ failure assessment (SOFA) score from baseline in patients with confirmed diagnosis of systemic anthrax treated with AIGIV. Total SOFA score can range from 0 to 24; increase in total SOFA score suggests worse clinical outcome prediction.
Assessment of AIGIV pharmacokinetics | Up to Day 7
  Serum concentration of AIGIV over time in patients with confirmed diagnosis of systemic anthrax treated with AIGIV to determine pharmacokinetic parameters such as maximum serum concentration, area under the concentration versus time (i.e. level of AIGIV circulating over time) and clearance
Assessment of anthrax toxin levels (protective antigen and lethal factor) | Up to Day 7
  Levels of anthrax toxins (protective antigen and lethal factor) over time in patients with confirmed diagnosis of systemic anthrax treated with AIGIV

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Essink, MD, Principal Investigator